CLINICAL TRIAL: NCT06088914
Title: Behavioral and Neural Correlates of Post-Stroke Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-FY2023-226; 1R15HD109737-01A1 (NIH); R15HD109737 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-10-18 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Fatigue
MeSH Terms: conditions — Stroke; Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Anodal tDCS group (Experimental): Participants will receive anodal tDCS applied to the ipsilesional primary motor cortex.
  Interventions: Device: Anodal transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Participants will receive sham tDCS applied to the ipsilesional primary motor cortex
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation — Anodal tDCS will be delivered for 5 consecutive days. Participants will receive 2 mA of stimulation for 20 minutes with the anodal electrode placed on the ipsilesional primary motor cortex (M1) and the cathodal electrode placed over the contralateral supraorbital area.
  Arms: Anodal tDCS group
Device: Sham transcranial direct current stimulation — Sham tDCS will be delivered for 5 consecutive days. Participants will receive sham stimulation for 20 minutes with the current intensity ramping down after 30 seconds of stimulation. The anodal electrode placed on the ipsilesional primary motor cortex (M1) and the cathodal electrode placed over the contralateral supraorbital area.
  Arms: Sham tDCS

SUMMARY:
The goal of this phase I/II clinical trial is to determine the behavioral and neural effects of 5-daily transcranial direct current stimulation on post-stroke fatigue. The three aims are:

Aim 1: Investigate the behavioral effect of 5 daily sessions of anodal tDCS over the ipsilesional M1 on PSF.

Aim 2: Investigate the neurophysiological effect of 5 daily sessions of anodal tDCS over the ipsilesional M1.

Aim 3: Determine the relationship between changes in M1 excitability, brain connectivity and changes in PSF.

Participants will receive either a real or sham stimulation for 5 consecutive days and fatigue will be assessed before, immediately after and 1-month after the intervention. Fatigue will be assessed using clinical, behavioral, and neurophysiological outcomes.

DETAILED DESCRIPTION:
Up to 85% stroke survivors experience post-stroke fatigue (PSF) defined as intensified perceived effort during activities. PSF is a significant barrier to full participation in rehabilitation and negatively affects quality of life after stroke. Despite its well-known impacts, there are very few targeted interventions for PSF largely due to unclear underlying mechanisms. A few brain stimulation studies have suggested a relationship between primary motor cortex (M1) excitability and PSF. Recent clinical trials using anodal transcranial direct current stimulation (tDCS) to modulate brain excitability reported mixed clinical efficacy in reducing PSF with unclear mechanisms of action.

The proposed research will address the gaps in our knowledge by determining the behavioral and neural correlates of PSF using an experimental design and multimodal approach.

Thirty-two individuals with significant fatigue due stroke will be randomly assigned to receive five consecutive sessions of anodal or sham tDCS. Before and after intervention, participants will complete clinical and behavioral assessments of PSF, brain excitability assessment using transcranial magnetic stimulation, and brain connectivity assessment using resting state functional MRI. In aim 1, the investigators will determine if upregulating M1 excitability via tDCS will reduce PSF assessed by clinical and behavioral markers. Aim 2 will utilize brain stimulation and brain imaging techniques to probe the neurophysiological effect of tDCS on PSF. Aim 3 will explore the relationship between changes in neurophysiological outcomes and changes in PSF.

The long-term goal of the team is to develop evidence based, theory-driven interventions to manage PSF. The proposed study is innovative in that it investigates a relative novel intervention to mitigate PSF and adopts a multimodal approach to examine the underlying mechanisms. The comprehensive research will guide the development of treatment targeted the underlying mechanisms of PSF. In addition to its scientific and clinical significances, the proposed research will achieve its educational goals by fostering a group of student researchers and promoting rigorous research cultures within the investigator's institute.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years old;
2. have a history of unilateral stroke ≥ 3 months prior to enrollment to ensure stability;
3. have an average score ≥ 4 on FSS;
4. have some movement capability in the more affected arm (upper extremity Fugl-Meyer(FMUE) ≥ 28) to ensure they can perform the reaching task;
5. be able to follow three-step commands.

Exclusion Criteria:

1. acute medical problems;
2. the presence of any contraindication to tDCS, MRI or TMS;
3. the presence of significant depression (score > 10 on the Patient Health Questionnaire-9);
4. significant pain in the upper extremities that interferes with movements; or
5. use of medication which may affect the level of fatigue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale score | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  This is a 9 item questionnaire and each item is rated on a Likert scale 1-7. Participants will rate their responseS based on their previous week experience. A higher score suggests more fatigue.
Input-output curve slope | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Brain excitability will be indexed using the input-output curve slope acquired with single-pulse transcranial magnetic stimulation (TMS)protocol. A greater slope value indicates a greater brain excitability.

SECONDARY OUTCOMES:
Borg Rating of Perceived Exertion | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Participants will rate their perceived physical effort associated with a reaching task on a scale ranging from 6 to 20. A higher rating suggests higher perceived effort.
Functional connectivity of the fronto-striato-thalamic network | This outcome will be assessed at 2 time points during the study, at baseline and immediately after the intervention ( an average of 7 days from baseline).
  Brain functional connectivity will be evaluated using 10-minute resting state functional MRI. A greater correlation coefficient value indicates a greater connectivity within the network.
Fatigue Scale for Motor and Cognitive Function | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  This is a 20-item questionnaire and each item is rated on a 5-point Likert scale. The questionnaire yields one motor and one cognitive scores. A higher score indicates more fatigue.
Visual Analog Scale-Fatigue | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  This is a 10cm single dimension scale with a higher score indicates a higher level of fatigue.
Paas Mental Effort Rating Scale | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Participants will rate their perceived mental effort associated with a reaching task on a scale ranging from 1 to 9. A higher score indicates greater mental effort perceived.
Paired pulse Transcranial Magnetic Stimulation measures | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Brain excitability will also be indexed using neurophysiological measures acquired with paired pulse transcranial magnetic stimulation protocol. These include short-interval intracortical inhibition (SICI) and intracortical facilitation (ICF).

OTHER OUTCOMES:
Functional connectivity of other established brain networks. | This outcome will be assessed at 2 time points during the study, at baseline and immediately after the intervention ( an average of 7 days from baseline).
  Using the 10-minute resting state functional MRI data acquired, the functional connectivity of other established networks, including sensorimotor network, fronto-parietal network, and default mode network will be explored.
Reach movement time | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Movement time (measured in seconds) will be used to index reach performance with a shorter movement time indicating a better performance.
Reach reaction time | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Reaction time (measured in seconds) will be used to index reach planning with a shorter reaction indicating a better performance.
Reach error | This outcome will be assessed at 3 time points during the study, at baseline, immediately after the intervention ( an average of 7 days from baseline) and at follow-up (an average of 5 weeks from baseline)
  Error (measured in cm) will be used to index movement accuracy with a lower error indicating a better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ting Goh, Principal Investigator — Physical Therapy
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the manuscripts, the de-identified data generated from the project will be made available to qualified researchers outside our research team upon request.
  The investigators will also deposit the de-identified data to the NICHD Data and Specimen Hub (DASH).
Supporting Information: Study Protocol
Time Frame: Upon the publication of the manuscripts (~12 months after study completion).
Access Criteria: Qualified researchers can contact PI via email (hgoh1@twu.edu) to request access to the de-identified data.
  DASH users can request access to the de-identified data deposited to the NICH DASH.

REFERENCES:
- [Derived] Liao KC, Christian I, Stewart J, Trudelle-Jackson E, Wang W, Shang T, Goh HT. Behavioral and Neural correlates of Post-STROKE Fatigue: A randomized controlled trial protocol. PLoS One. 2025 Jun 6;20(6):e0324591. doi: 10.1371/journal.pone.0324591. eCollection 2025. PMID 40478794